CLINICAL TRIAL: NCT00954031
Title: Impact of Anti-inflammatory and Antibiotic Therapy on the Emergence of Peri-tonsillar Abscess
Acronym: APA
Status: Terminated | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: General director, Nantes University Hospital
Other Study IDs: BRD 08/9-W
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Abscess, Peritonsillar
MeSH Terms: conditions — Peritonsillar Abscess

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- case: hospitalized patients, adult or child, including the diagnosis of APA was made, after consulting their physician.
- The control group: Two patients witnesses will be matched to each case:
  Chronological criterion: consultation for a "sore throat" 10 days (± 3 days) before the date of hospitalization of cases, between 13 and J-J-7.
  Age criteria: year of birth ± 5 years Geographical criteria: living in the same department, failing in an adjacent Department Social criteria: beneficiary or otherwise of the CMU, to avoid a selection bias leading social most frequently at the onset of the APA

SUMMARY:
Analyze in children and adults, risk factors in the onset of the APA. The main hypothesis focuses on the use of anti-inflammatory in the context of pharyngitis or sore throat before the symptoms of ABS. Secondary objectives:

1. - Analyze the implementation of a rapid diagnostic test and its result on the occurrence of an ABS
2. - Measure the frequency of prescription and describe the reasons for not prescribing an antibiotic for patients who consulted for a sore throat and having developed a PLA
3. - Describe the microbial flora could puncture of patients hospitalized for APA

ELIGIBILITY:
Inclusion Criteria:

* clinical existence of a PLA (phlegmon), validated by a senior ENT, usually (but not necessarily) following a request by an emergency. The visible appearance to the merits throat must justify puncture. Cases will be included whether or not they had consulted for a "sore throat" in the 10 days preceding the date of diagnosis

Exclusion Criteria:

* Neoplastic disease of the throat, scalable Hematologic with tonsillar localization History of tonsillectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients, adult or child, including the diagnosis of APA was made, after consulting their physician
Sampling Method: Non-Probability Sample
Enrollment: 711 (Estimated)
Dates: Start 2009-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The principal judgement criterion of the study is the positive diagnosis of an APA. The explanatory variables to meet the main objective is the drug exposure (anti-inflammatory) | 2,5 years

SECONDARY OUTCOMES:
The explanatory variables to meet the secondary objectives are: - The creation of a TDR - The prescription of antibiotics - The diagnosis of angina Strep Group A - The identification of a group A streptococcus in t | 2,5 years

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Potel, PhD, Principal Investigator — Nantes University Hospital
Locations (15):
- France (15):
  - Nantes University Hospital, Nantes, Pays de Loire
  - Angers university Hospital, Angers
  - Caen universty Hospital, Caen
  - Clermont Ferrand University Hospital, Clermont-Ferrand
  - Grenoble University Hospital, Grenoble
  - Lille University Hospital, Lille
  - Ambroise Paré Hospital, Paris
  - Paris-Bichat-Hospital, Paris
  - Paris-Cochin Hospital, Paris
  - Paris-Lariboisière Hospital, Paris
  - Paris-Tenon-Hospital, Paris
  - Poitiers University Hospital, Poitiers
  - Rennes University hospital, Rennes
  - Toulouse University Hospital, Toulouse
  - Tours University Hosipital, Tours